CLINICAL TRIAL: NCT05076370
Title: Cannabidiol Pharmacotherapy for Comorbid Opioid Addiction and Chronic Pain
Brief Title: Safety and Tolerability of Cannabidiol Among Persons With Opioid Use Disorder Receiving Methadone or Buprenorphine
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Joao De Aquino, Principal Investigator, Yale University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2000029286; 1K23DA052682-01 (NIH)
Record Dates: First submitted 2021-09-29; First posted 2021-10-13 (Actual); Results first posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-10

CONDITIONS: Addiction
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Intervention Model Description: Initial safety pilot phase of 6 participants,(3 methadone and 3 on Buprenorphine) The general study is a randomized, placebo-controlled, crossover human laboratory study investigating the dose-dependent safety and acute effects of CBD on measures of pain and opioid craving in outpatients with OUD receiving methadone or buprenorphine.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CBD 400mg (Active Comparator): CBD 400mg
  Interventions: Drug: CBD Day 1
- CBD 800mg (Active Comparator): CBD 800mg
  Interventions: Drug: CBD Day 2
- CBD 1200mg (Active Comparator): CBD 1200mg
  Interventions: Drug: CBD Day 3

INTERVENTIONS:
Drug: CBD Day 1 — CBD 400mg
  Arms: CBD 400mg
Drug: CBD Day 2 — CBD 800mg
  Arms: CBD 800mg
Drug: CBD Day 3 — CBD 1200mg
  Arms: CBD 1200mg

SUMMARY:
The overarching goal of this study is to evaluate the potential of Cannabidiol (CBD) as an adjunctive treatment for comorbid opioid use disorder (OUD) and chronic pain. This is a randomized, placebo-controlled, crossover human laboratory study investigating the dose-dependent safety and acute effects of CBD on measures of pain and opioid craving in outpatients with OUD receiving methadone or buprenorphine.

DETAILED DESCRIPTION:
An initial safety pilot phase will recruit six participants: three receiving treatment with methadone and three receiving treatment with buprenorphine. If the results of the pilot study support the safety of CBD administration in this clinical sample, the general study will recruit participants with comorbid OUD and chronic pain, with half the subjects receiving methadone and half receiving buprenorphine. Both sub-studies will enroll participants who do not currently require an inpatient hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 70 years old.
* Diagnosed with OUD and currently enrolled in methadone or buprenorphine maintenance treatment.
* Having chronic pain, uniformly operationalized as grade II (high-intensity) non- cancer pain for ≥ 6 months 49.
* Capable of providing informed consent in English.
* Compliant in opioid maintenance treatment and on a stable dose for four weeks or longer.
* Not meeting DSM-5 criteria for substance use disorders other than OUD or tobacco use disorder within the last 12 months.
* No current medical problems deemed contraindicated for participation by principal investigator.
* For women, not pregnant as determined by pregnancy screening; not breast-feeding; using acceptable birth control methods. Acceptable contraception for women includes oral contraceptives, contraceptive depot injections, contraceptive subdermal implants, intrauterine devices, or surgical contraception methods. Acceptable contraception for men includes condoms or surgical contraception methods.

Exclusion Criteria:

* Other current major psychiatric disorders deemed clinically unstable by the principal investigator, such as severe depression and/or active suicidal ideation.
* Having experienced major psychosocial stressors recently (≤ 6 weeks before enrollment), at the discretion of the principal investigator.
* Methadone dose under 60mg or over 100mg
* Buprenorphine over 24mg.
* Having received inpatient psychiatric treatment recently (≤ 60 days before enrollment).
* Candidates receiving products containing either THC or CBD will be excluded.
* Current use regular use other prescription opioids, gabapentinoids (pregabalin, gabapentin), antidepressants (SSRIs, SNRIs, TCAs), benzodiazepines, platelet inhibitors (e.g., clopidogrel, apixaban, ticagrelor), or NSAIDs.
* Current weight of less of 60 kg.
* Allergy to sesame seed oil, which is an ingredient of the CBD formulation used.
* Serious medical or neurological illness or treatment for a medical disorder that could interfere with study participation as determined by principal investigator.
* Participants who have elevation of liver enzymes (ALT and/or AST) 2x above the normal limit or higher.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joao De Aquino, M.D., Principal Investigator — Yale University
Locations (1):
- Veteran Affairs Hospital, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through responses to fliers, craigslist, clinicaltrials.gov, BuildClinical and through local mental health and substance use disorder treatment facilities
Groups:
- CBD Overall: Using a dose-escalation paradigm, crossover assignment, participants were administered single doses of 400 mg, 800 mg, and 1200 mg of CBD, across 3 test sessions.
Period: Overall Study
Arm/Group | CBD Overall
Started | 7
Completed 400mg CBD | 7
Completed 800mg CBD | 7
Completed 1200mg CBD | 6
Receiving Methadone | 4
Receiving Buprenorphine | 3
Completed | 6
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Per protocol population. Defined as participants completing the experimental drug conditions.
Groups:
- Buprenorphine: Completers (3 receiving buprenorphine)
- Methadone: Completers (4 receiving methadone)
- Total: Total of all reporting groups
Arm/Group | Buprenorphine | Methadone | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (2) | 40 (2.3) | 40 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 7
Buprenorphine or Methadone Dose [Mean (Standard Deviation); unit: milligrams] — Population: Participants received buprenorphine or methadone.
  milligrams
    Buprenorphine: number analyzed (Participants) | 3 | 0 | 3
    Buprenorphine | 11.3 (2.4) |  | 11.3 (2.4)
    Methadone: number analyzed (Participants) | 0 | 4 | 4
    Methadone |  | 91.2 (5.2) | 91.2 (5.2)
Weight [Mean (Standard Deviation); unit: Pounds (lbs)] | 193.3 (20.5) | 223.8 (28.7) | 210.7 (18.2)
Brief Pain Index (BPI) [Mean (Standard Deviation); unit: score on a scale] — The BPI Severity and Interference each have a total score range of 0-10 where: 0 = no pain, 1-3 = mild pain, 4-6 = moderate pain, 7-10 = severe pain.
  score on a scale
    Severity | 5.3 (1.4) | 1.7 (2.6) | 3.2 (2.8)
    Interference | 5.7 (2.2) | 1.5 (2.4) | 3.3 (3.1)
Clinical Pain Location [Count of Participants; unit: Participants]
  Back | 3 | 1 | 4
  Knee | 2 | 1 | 3
  Neck | 1 | 1 | 2
  Shoulder | 1 | 1 | 2
  Other | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Agitation Calmness Evaluation Scale (ACES)
Description: The ACES consists of a single item that rates overall agitation and sedation of the participant at the time of evaluation, where 1 indicates marked agitation; 2: moderate agitation; 3: mild agitation; 4: normal behavior; 5: mild calmness; 6: moderate calmness; 7: marked calmness; 8: deep sleep; and 9: unarousable. Clinically significant sedation was a priori defined as an ACES score of 7 (marked calmness) or higher at any point during the session. A score was averaged across all time intervals.
Time Frame: Baseline (30 minutes before the administration of CBD), hourly for 4 hours after the administration of methadone (administered +210 minutes after CBD) and 3 hours after the administration of buprenorphine (administered +210 minutes after CBD)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBD 400mg | CBD 800mg | CBD 1200mg
Number analyzed (Participants) | 7 | 7 | 7
score on a scale
  Baseline (-30 Minutes) | 4 (0) | 4 (0) | 4 (0)
  +270 Minutes | 4.07 (0.40) | 4 (0) | 4.01 (0.11)
  +330 Minutes | 4.02 (0.24) | 4 (0) | 4 (0)
  +390 Minutes | 4 (0) | 4 (0) | 4 (0)
  +450 Minutes | 4 (0) | 4 (0) | 4 (0)

2. Primary Outcome: Mini Mental Status Examination (MMSE)
Description: The MMSE is a 30-point scale ranging from 0 to 30 that measures five areas of cognitive function: orientation, registration, attention and calculation, recall, and language. Each scale is summed to compute a total score. The MMSE is used extensively in clinical and research settings to measure cognitive impairment. A score of 24 or higher is generally considered within the normal range, while lower scores suggest potential cognitive impairment. Scores are often interpreted as follows: 25-30 = normal cognition, 21-24 = mild impairment, 10-20 = moderate impairment, and below 10 = severe impairment.
Time Frame: Baseline (30 minutes before the administration of CBD), hourly for 4 hours after the administration of methadone (administered +210 after CBD) and 3 hours after the administration of buprenorphine (administered +210 minutes after CBD)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBD 400mg | CBD 800mg | CBD 1200mg
Number analyzed (Participants) | 7 | 7 | 7
score on a scale
  Baseline (-30 minutes) | 29.43 (0.98) | 29.33 (1.21) | 29.50 (0.55)
  +270 Minutes | 29.86 (0.38) | 29.33 (0.82) | 29.83 (0.41)
  +330 Minutes | 29.57 (0.79) | 29.57 (0.53) | 29.14 (1.46)
  +390 Minutes | 30 (0) | 29.33 (1.03) | 29.43 (0.53)
  +450 Minutes | 29.50 (0.58) | 29.50 (0.58) | 29.67 (0.58)

3. Primary Outcome: Systematic Assessment of Side Effects (SAFTEE)
Description: The SAFTEE is a multi-symptom checklist that has been used successfully in our previous studies to assess and monitor any adverse events and possible side effects of study medications. It includes information regarding the severity of any presenting symptoms (0= none, 1= mild, 2= moderate, and 3= severe), as well as the course of action taken by the study staff in response. The SAFTEE was administered before the administration of CBD at baseline, (timepoint -30 minutes) and 4.5 hours after the administration of CBD (timepoint +240 minutes) during each test session. Data presented here is the number of participants that reported symptoms on SAFTEE.
Time Frame: baseline and 4.5 hours after the administration of CBD
Measure: Count of Participants; unit: Participants
Arm/Group | CBD 400mg | CBD 800mg | CBD 1200mg
Number analyzed (Participants) | 7 | 7 | 7
Participants | 5 | 5 | 5

4. Secondary Outcome: Quantitative Sensory Testing (QST)- Threshold and Tolerance
Description: Pain threshold and tolerance will be assessed using a comprehensive QST battery. This is a reliable, dynamic, and computerized method of quantifying distinct mechanisms of the pain experience. QST measures are sensitive to the effects of cannabinoids, important biomarkers of chronic pain, and predictors of the pain treatment response. Threshold: the temperature the participant first begins to feel pain (average pain threshold), and when the participant can no longer tolerate the stimuli (Tolerance). The temperature ranges from 37 degrees celsius to 50 degrees celsius. A lower temperature represents a lower pain threshold and a higher temperature represents a higher pain threshold. A lower temperature represents a lower pain tolerance and a higher temperature represents a higher pain tolerance.
Time Frame: baseline, 2 hours and 4 hours after the administration of CBD.
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | CBD 400mg | CBD 800mg | CBD 1200mg
Number analyzed (Participants) | 7 | 7 | 7
degrees Celsius
  Threshold Baseline | 40.29 (5.6) | 40.55 (4.3) | 41.435 (4.36)
  Threshold 2 hours | 39.65 (3.85) | 40.47 (4.27) | 40.63 (4.3)
  Threshold 4 hours | 39.95 (3.99) | 40.47 (3.9) | 39.94 (4.33)
  Tolerance Baseline | 46.17 (3.57) | 46.33 (3.4) | 47.08 (2.76)
  Tolerance 2 hours | 46.70 (2.66) | 45.82 (3.9) | 45.07 (4.35)
  Tolerance 4 hours | 45.74 (3.62) | 46.66 (2.86) | 45.81 (3.88)

5. Secondary Outcome: Change in Quantitative Sensory Testing (QST) Conditioned Pain Modulation (CPM)
Description: CPM indexes top-down pain inhibition, by leveraging the "pain inhibits pain phenomena". In CPM, a test stimulus is rated on a -100 to +100 Numeric Rating Scale (NRS) for pain both alone and during a concurrent conditioning stimulus applied elsewhere on the body. The CPM Score is the difference between these two ratings.
  CPM score is a Difference (Delta): Pain rating (test stimulus alone) - Pain rating (test stimulus with conditioning stimulus) Interpretation: Higher (more positive) values indicate greater pain inhibition.
Time Frame: Baseline (-30 minutes), 2 hours (+120 minutes), and 4 hours (+240 minutes) after the administration of CBD.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBD 400mg | CBD 800mg | CBD 1200mg
Number analyzed (Participants) | 7 | 7 | 7
units on a scale
  Baseline (-30 Minutes) | 3.43 (11.69) | 5.29 (12.4) | 5.7 (5.6)
  +120 Minutes | 2.14 (5.81) | -4.28 (6.21) | 1.71 (2.98)
  +240 Minutes | -9.86 (22.99) | -6.28 (10.17) | -4.42 (11.88)

6. Secondary Outcome: Quantitative Sensory Testing (QST) Temporal Summation of Pain (TSP)
Description: Pain will be assessed using a comprehensive QST battery. QST measures are sensitive to the effects of cannabinoids, important biomarkers of chronic pain, and predictors of the pain treatment response. TSP involves the repeated administration of noxious stimuli, indexing bottom-up pain facilitation. Therefore, TSP measures the increase in pain perception with repeated noxious stimuli, calculated as the area under the curve (AUC) of pain ratings over time during repeated stimulation.
  Higher TSP scores indicate worse outcomes (greater pain facilitation/central sensitization), while lower TSP scores indicate better outcomes (less pain facilitation/central sensitization). The TSP AUC values represent the cumulative pain experience during repeated stimulation (VAS units*seconds), where larger values reflect greater temporal summation of pain, which is associated with central nervous system sensitization and chronic pain conditions.
Time Frame: Baseline, 2 hours and 4 hours after the administration of CBD.
Measure: Mean (Standard Deviation); unit: AUC (VAS units*seconds)
Arm/Group | CBD 400mg | CBD 800mg | CBD 1200mg
Number analyzed (Participants) | 7 | 7 | 7
AUC (VAS units*seconds)
  Baseline (-30 Minutes) | 522436.5 (784227.4) | 333689.75 (596722.19) | 337314.16 (641890.80)
  +120 Minutes | 549573 (841674.11) | 354263.75 (693645.10) | 390454.3 (670332.51)
  +240 Minutes | 445697.91 (697669.30) | 260961.4 (399847.43) | 542224.7 (731050.04)

7. Other Pre Specified Outcome: Change in The Heroin Craving Questionnaire - Short Form 14 (HCQ-SF-14)
Description: The Heroin Craving Questionnaire - Short Form 14 (HCQ-SF-14) consists of 14 statements about the respondent's feelings and thoughts about using heroin as he or she is completing the questionnaire (i.e., right now). Each of the 14 items is scored on a scale from 1 (Strongly Disagree) to 7 (Strongly Agree). The HCQ-SF-14 score is obtained by adding the scores of all 14 statements and dividing the total by 14. Higher scores on the HCQ-SF-14 indicate a stronger craving for heroin.
  The HCQ-14 was administered before (+150 minutes) and after (+155 minutes) participants watched a cue-induced craving video. The difference of the two HCQ-14 scores (post - pre) will be used to index cue-elicited craving.
Time Frame: Average difference of scores from before cue-induced craving video (+150 minutes) and after cue-induced craving video (+155 minutes)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- CBD 400mg: CBD 400mg CBD Day 1: CBD 400mg
- CBD 800mg: CBD 800mg CBD Day 2: CBD 800mg
- CBD 1200mg: CBD 1200mg CBD Day 3: CBD 1200mg
Arm/Group | CBD 400mg | CBD 800mg | CBD 1200mg
Number analyzed (Participants) | 7 | 7 | 7
units on a scale | -0.57 (3.05) | -0.56 (3.69) | 0.33 (2.58)

ADVERSE EVENTS:
Time Frame: baseline up to 6 hours post CBD
Arm/Group | CBD 400mg | CBD 800mg | CBD 1200mg
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 1/7
Other Adverse Events (participants affected / at risk) | 5/7 | 6/7 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CBD 400mg (N=7) | CBD 800mg (N=7) | CBD 1200mg (N=7)
Unrelated Serious Adverse Event (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CBD 400mg (N=7) | CBD 800mg (N=7) | CBD 1200mg (N=7)
Agitation (General disorders) | 0 | 0 | 1
Anger or irritability (General disorders) | 0 | 0 | 1
Back, muscle or bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Chest pain (Cardiac disorders) | 0 | 0 | 1
Chills (General disorders) | 0 | 1 | 0
Confusion (General disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 3 | 2
Depressed mood (Psychiatric disorders) | 2 | 2 | 1
Difficulty concentrating (General disorders) | 0 | 0 | 1
Dry mouth (General disorders) | 0 | 0 | 2
Excessive hunger (General disorders) | 1 | 0 | 0
Extreme thirst (General disorders) | 1 | 1 | 1
Feeling dizzy or faint or lightheaded (General disorders) | 0 | 0 | 1
Feeling Drowsy (General disorders) | 4 | 4 | 4
Headache (General disorders) | 1 | 2 | 1
Heartburn (Metabolism and nutrition disorders) | 1 | 2 | 1
Irregular or pounding heartbeat (Cardiac disorders) | 0 | 0 | 1
Loss of appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Memory problems (General disorders) | 0 | 0 | 1
Mood swings (Psychiatric disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Nervousness (General disorders) | 1 | 2 | 1
Problems with urination (General disorders) | 0 | 2 | 0
Restlessness (General disorders) | 2 | 2 | 1
Runny nose (General disorders) | 1 | 3 | 1
Stomach pain (Gastrointestinal disorders) | 1 | 0 | 1
Sweating (General disorders) | 0 | 2 | 1
Teary or dry eyes (General disorders) | 0 | 0 | 2
Tremors or shakiness (General disorders) | 0 | 0 | 1
Trouble walking (General disorders) | 0 | 0 | 1
Upset stomach (Gastrointestinal disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-05): https://cdn.clinicaltrials.gov/large-docs/70/NCT05076370/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/70/NCT05076370/ICF_001.pdf